CLINICAL TRIAL: NCT01905644
Title: Verifying Anal Sphincter Integrity in the Delivery Room Using a Specific Perineal Ultrasound: Impact on Immediate Care and Postpartum Anal Incontinence Rates in Mothers Undergoing Vaginal Birth
Brief Title: Verifying Post-delivery Anal Sphincter Integrity Using Perineal Ultrasound: Impact on Immediate Care
Acronym: OASIS 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AOI/2012/VL-01; 2013-A00773-42 (Other: RBC number)
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Delivery, Obstetric
Keywords: Vaginal delivery; Perineal lesions; Anal sphincter rupture; Ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With ultrasound (Experimental): Patients in this group will have perineal ultrasound for the detection of anal sphincter ruptures.
  Intervention: Perineal ultrasound
  Interventions: Procedure: Perineal ultrasound
- Without ultrasound (No Intervention): Patients in this group will not have perineal ultrasound for the detection of anal sphincter ruptures.

INTERVENTIONS:
Procedure: Perineal ultrasound — Perineal ultrasound will be used after delivery to help detect anal sphincter ruptures.
  Arms: With ultrasound

SUMMARY:
The main objective of this study is to compare post partum rates of anal sphincter rupture (that is to say the rate of sutures) diagnosed in women with ≥ 2nd degree vaginal tears between two groups: (1) women who are screened just after delivery by performing a perineal ultrasound versus a similar group of women who did not receive screening. This study was not designed to evaluate ultrasound as a diagnostic test but to compare the rate of perineal surgical procedures in each arm.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. Compare the anal incontinence score (measured by the Wexner score, qualitative and quantitative assessment) at 3 months between the two groups.

B. To assess the safety of perineal ultrasound in the group with "ultrasound" using a visual analog scale for discomfort

C. Assess the inter and intra operator consistency of perineal ultrasound snapshot readings

D. Evaluate and compare the rate of infectious complications of perineal sutures between the two groups at 3 months.

E. Evaluate and compare the quality of life (questionnaires PFIQ, PFDI, SF36, Euroqol) between the two groups at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 3 months of follow-up
* Paturient, vaginal births only
* Presence of >= stage 2 perineal lesion
* Patient accepts a priori the performance of a perineal ultrasound

Exclusion Criteria:

* The patient is participating in another study (excepting BBBOX (2011-A00327-36), ElastoMAP (2013-A01148-37), ElastoDéclench, BAKRI, Papillo PMA, GrossPath, LXRs, DGPostPartum, "scalp lactates", and UpSideDown studies)
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* Delivery by C-section
* Intact perineum after delivery (no indication for perineal surgery in light of absence of vaginal lesion)
* Emergency situation preventing time for perineal ultrasound
* History of anal incontinence before giving birth
* Allergy to ultrasound gel

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2014-03-07 (Actual); Primary Completion 2016-11-24 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Presence/absence of an anal sphincter rupture | Day 0

SECONDARY OUTCOMES:
Wexner score for anal incontinence | Day 0
Wexner score for anal incontinence | 3 months
Tolerance of perineal ultrasound | Day 0
  Visual analog scale (0 to 10) used to evaluate discomfort.
Kappa coefficient for inter-operator ultrasound reading | Day 0
Kappa coefficient for intra-operator ultrasound reading | Day 0
Presence/absence of suture infection | 3 months
PFIQ questionnaire | Day 0
PFIQ questionnaire | 3 months
PFDI questionnaire | Day 0
PFDI questionnaire | 3 months
SF36 questionnaire | Day 0
SF36 questionnaire | 3 months
Euroqol questionnaire | Day 0
Euroqol questionnaire | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Letouzey, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - CHU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CHU de Poitiers, Poitiers